CLINICAL TRIAL: NCT03720717
Title: Baclofen as a Perioperative Analgesic Adjuvant
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Futility analysis at midpoint analysis
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Timothy Ness, MD, Prinicipal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300002466
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Baclofen

STUDY DESIGN:
Intervention Model Description: Coded envelopes with study drug/placebo had been generated and randomized. Patients were enrolled and given drug in next envelope. After completion of study patients assigned into opioid-naive or daily opioid-tolerant groups based on history given by patient
Who Masked: Participant, Care Provider
Masking Description: Coded envelopes as described above
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Opioid Tolerant - baclofen (Experimental): Patients identified as opioid tolerant if they reported using daily opioids greater than one month. Randomized into baclofen (10 mg p.o.) group. Drug was given within 30 minutes of OR entry. Although pseudo-randomization was planned to be initiated near the end of the trial in order to assure balance group numbers, the early termination of the study did not require this and so all randomized to either baclofen or placebo, independent of opioid status.
  Interventions: Drug: Baclofen 10mg
- Opioid Tolerant - placebo (Placebo Comparator): Patients identified as opioid tolerant if they reported using daily opioids greater than one month. Randomized into placebo group with dummy pill administration. Pill was given within 30 minutes of OR entry.Although pseudo-randomization was planned to be initiated near the end of the trial in order to assure balance group numbers, the early termination of the study did not require this and so all randomized to either baclofen or placebo, independent of opioid status.
  Interventions: Other: Placebo
- Opioid Naive - baclofen (Experimental): Patients identified as opioid naive if they reported minimal preoperative use of opioids with a criteria of non-daily use and/or use less than one month. Randomized into baclofen (10 mg p.o.) group. Drug was given within 30 minutes of OR entry.Although pseudo-randomization was planned to be initiated near the end of the trial in order to assure balance group numbers, the early termination of the study did not require this and so all randomized to either baclofen or placebo, independent of opioid status.
  Interventions: Drug: Baclofen 10mg
- Opioid Naive - placebo (Placebo Comparator): Patients identified as opioid naive if they reported minimal preoperative use of opioids with a criteria of non-daily use and/or use less than one month. Randomized into placebo group with dummy pill administration. Pill was given within 30 minutes of OR entry.Although pseudo-randomization was planned to be initiated near the end of the trial in order to assure balance group numbers, the early termination of the study did not require this and so all randomized to either baclofen or placebo, independent of opioid status.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Baclofen 10mg — Baclofen administration pre-operatively
  Other Names: Lioresol
  Arms: Opioid Naive - baclofen; Opioid Tolerant - baclofen
Other: Placebo — Placebo administration
  Arms: Opioid Naive - placebo; Opioid Tolerant - placebo

SUMMARY:
The purpose of this study is to determine whether a single, oral dose of baclofen alters postoperative opioid requirements.

DETAILED DESCRIPTION:
Postoperative pain continues to be a significant clinical problem. Use of perioperative adjuvants has improved postoperative pain control. The GABA-B receptor agonist, baclofen, is an appropriate drug to trial as such an analgesic adjuvant. Therefore, the investigators will conduct a study designed to determine whether or not a single, oral dose of baclofen given to patients undergoing kidney stone surgery will reduce postoperative opioid requirements measured in the first 24 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >= 19 y.o.) scheduled for kidney stone-related surgery

Exclusion Criteria: (note - there were no patients requiring exclusion)

* History of allergy to baclofen
* Any condition which might limit appropriate report and treatment of postoperative pain (e.g., non-English speaking; severe psychiatric disease)
* Active history of cancer
* Potential for difficult airway as judged by attending anesthesiologist due to concerns there could be muscle weakness from the drug with consequent respiratory depression

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mandabach, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data available on reasonable request - currently in RedCap system
Supporting Information: CSR
Time Frame: Published - Cureus 2024 - DOI: 10.7759/cureus
Access Criteria: published

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opioid Tolerant - Baclofen | Opioid Tolerant - Placebo | Opioid Naive - Baclofen | Opioid Naive - Placebo
Started (Enrollment for all four groups of the study started on October 27, 2020. Study occurred during a single 24 hour period. Code was broken at midpoint analysis identifying specific groups) | 5 | 7 | 12 | 10
Completed | 5 | 7 | 12 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid Tolerant - Baclofen | Opioid Tolerant - Placebo | Opioid Naive - Baclofen | Opioid Naive - Placebo | Total
Number analyzed (Participants) | 5 | 7 | 12 | 10 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11 | 8 | 30
  >=65 years | 0 | 1 | 1 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (11.6) | 45.3 (17.0) | 51.5 (16.6) | 46.6 (19.4) | 49.7 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 5 | 3 | 16
  Male | 0 | 4 | 7 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 7 | 12 | 10 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 2 | 7
  White | 4 | 5 | 10 | 8 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12 | 10 | 34
Opioid use - >=30 Oral morphine equivalents consumed per day [Count of Participants; unit: Participants] | 5 | 7 | 12 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Requirements
Description: Patients Patients' opioid requirements for acceptable pain control will be assessed based on the total oral morphine equivalent needed for post operative pain control.
Time Frame: From 0 hours post-operatively to 24 hours post-operatively
Population: patients were stratified according to preprocedure opioid use into Opioid Tolerant and Opioid Naive groups based on above stated criteria
Measure: Mean (Standard Error); unit: mg oral morphine equivatents in 24 hours
Arm/Group | Opioid Tolerant - Baclofen | Opioid Tolerant - Placebo | Opioid Naive - Baclofen | Opioid Naive - Placebo
Number analyzed (Participants) | 5 | 7 | 12 | 10
mg oral morphine equivatents in 24 hours | 85.5 (33.6) | 96.8 (17.1) | 69.9 (10.0) | 40.4 (11.7)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Opioid Tolerant - Baclofen | Opioid Tolerant - Placebo | Opioid Naive - Baclofen | Opioid Naive - Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT03720717/Prot_SAP_002.pdf
  • Informed Consent Form (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT03720717/ICF_004.pdf